CLINICAL TRIAL: NCT05620225
Title: A Multicenter, Randomized, Clinical Trial Comparing the Safety and Effectiveness of Axon Therapy and Conventional Medical Management (AT+CMM) for the Treatment of Painful Diabetic Neuropathy to Sham and Conventional Medical Management (Sham+CMM)
Brief Title: Axon Therapy and Conventional Medical Management for Painful Diabetic Neuropathy Compared to Sham and Conventional Medical Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuraLace Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NLM-004
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2023-08

CONDITIONS: Neuralgia; Neuropathic Pain; Painful Diabetic Neuropathy
Keywords: transcutaneous magnetic stimulation; axon therapy; peripheral neuropathic pain; diabetic neuropathy
MeSH Terms: conditions — Neuralgia; Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, double blinded, randomized, multi-center clinical trial in which up to 80 subjects diagnosed with painful diabetic neuropathy will be randomized 3:1 into one of two treatment groups:
  1. Axon Therapy plus CMM (AT+CMM)
  2. Sham plus CMM (Sham+CMM)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects and clinical study staff (with the sole exception of the Blinding Operator) will be blinded to study treatment.
  Steps for setting up the device are extremely similar whether the patient is in the Sham or Active groups. The following steps must be completed before the patient or the Operator have entered the room for their session. Please avoid any unnecessary interactions with the patient, Operator or any other Clinic personnel in the performance of these tasks.
  The primary security method for protecting the Blind is strict utilization of Medrio and the special permissions granted by the Sponsor for the conduct of Blinding and Unblinding subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Axon Therapy + CMM (Experimental): Subjects will be consented, screened, and then undergo a 7-day baseline assessment period. Subjects will be asked to record pain, numbness, and sleep scores via a twice daily electronic diary. Subjects who meet inclusion criteria, including diary compliance, will undergo an in-clinic baseline evaluation (Day 1), be randomized, and start their treatments.
  All subjects will return to the clinic for treatments as follows:
  ● Day 1 - 30: 6 treatments
  * Week 1: 3 treatments
  * Week 2-4: Weekly treatments
  All subjects will return to the clinic for follow-up assessment at Day 30 (± 5 days). At the Day 30 visits subjects will be asked if they want to participate in Phase 2 of the study.
  Interventions: Device: Axon Therapy and CMM
- Sham + CMM (Sham Comparator): Subjects will be consented, screened, and then undergo a 7-day baseline assessment period. Subjects will be asked to record pain, numbness, and sleep scores via a twice daily electronic diary. Subjects who meet inclusion criteria, including diary compliance, will undergo an in-clinic baseline evaluation (Day 1), be randomized, and start their treatments.
  All subjects will return to the clinic for treatments as follows:
  ● Day 1 - 30: 6 treatments
  * Week 1: 3 treatments
  * Week 2-4: Weekly treatments
  All subjects will return to the clinic for follow-up assessment at Day 30 (± 5 days). At the Day 30 visits subjects will be asked if they want to participate in Phase 2 of the study.
  Interventions: Device: Sham and CMM

INTERVENTIONS:
Device: Axon Therapy and CMM — transcutaneous magnetic stimulation (TMS)
  Arms: Axon Therapy + CMM
Device: Sham and CMM — Sham and CMM
  Arms: Sham + CMM

SUMMARY:
Compare Axon Therapy plus conventional medical management (CMM) to Sham plus CMM in reducing neuropathic pain in patients with painful diabetic neuropathy (PDM).

DETAILED DESCRIPTION:
This is a two-phase study.

Phase 1 is a double blinded, two-arm, randomized, multi-center clinical trial to assess 1-month efficacy as compared to a sham group. Up to approximately 80 subjects diagnosed with painful diabetic neuropathy will be randomized 3:1 into one of two treatment groups:

1. Axon Therapy plus CMM (AT+CMM)
2. Sham plus CMM (Sham+CMM)

Subjects will be consented, screened, and then undergo a 7-day baseline assessment period. Subjects will be asked to record pain, numbness, and sleep scores via a twice daily electronic diary. Subjects who meet inclusion criteria, including diary compliance, will undergo an in-clinic baseline evaluation (Day 1), be randomized, and start their treatments.

All subjects will return to the clinic for treatments as follows:

● Day 1 - 30: 6 treatments

* Week 1: 3 treatments
* Week 2-4: Weekly treatments

All subjects will return to the clinic for follow-up assessment at Day 30 (± 5 days). At the Day 30 visits subjects will be asked if they want to participate in Phase 2 of the study.

Phase 2 of the study is an unblinded, one-arm, multi-center trial to assess extended efficacy of the treatment. At Day 30, subjects will be unblinded and allowed to remain in the study for an additional 60 (AT+CMM) to 90 (ATx+CMM) days. Those in the Sham arm can choose to crossover to active treatment ( ATx+CMM).

Subjects in the AT+CMM arm will return to the clinic as follows:

* Month 2: Bi-weekly treatment
* Month 3: Treatments every 2-4 weeks
* Additional treatments to treat flare ups; defined as an episode of pain with a VAS 6.

Subjects in the ATx+CMM arm will return to the clinic as follows:

* Month 2: 6 treatments

  * Week 1: 3 treatments
  * Week 2-4: Weekly treatments
* Month 3: Bi-weekly treatment
* Month 4: Treatments every 2-4 weeks
* Additional treatments to treat flare ups; defined as an episode of pain with a VAS 6.

Subjects who do not choose to remain in the study will be monitored for 30 days for AEs and then they will exit the study. The subject's reason for exiting the study will be recorded.

In addition to in-clinic assessments and treatments, all subjects will complete an electronic twice daily diary through Day 30 of the study (Day 60 for ATx+CMM subjects). Subjects will receive weekly phone follow-up for diary reminders and to assess for the occurrence of adverse events. Weekly phone follow-up will occur only during weeks when the subject is not seen in the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the study.
2. Subject is willing and able to comply with scheduled visits, treatment plan, daily pain, and other study procedures subject is able and willing to complete twice daily electronic diary for up to 60 days.
3. Subject must be literate in English to fill out the study questionnaires.
4. Men or women of any race or ethnicity who are 18-85 years of age.
5. Subjects must not have a Body Mass Index >40.
6. Subject must have painful diabetic neuropathy (Type 2) present in the lower limbs for more than three months per medical history
7. Subject has a pain score ≥5 on VAS at Enrollment/Screening Visit.
8. Subject has completed at least one of the two daily pain diary entries on at least five days between the Enrollment/Screening Visit and Visit 1 with a mean pain score of ≥4 and <10 based on Daily VAS to be eligible for the study.
9. Subject is on a stable pain medication regimen or is not taking pain medications, as

Exclusion Criteria:

1. Subjects with neuropathic pain due to post-herpetic neuropathy, HIV, trigeminal neuralgia; subjects whose post- traumatic neuropathic pain is categorized as central (e.g., spinal cord injury) rather than peripheral.
2. Subjects with any other chronic or recurrent pain syndrome rated greater than "mild" on a mild-moderate-severe scale, or which the investigator judges may interfere with the patients ability to report their pain accurately.
3. Any disorder that may be confused with PDN, such as tarsal tunnel syndrome, sciatica, bunions, ischemic claudication or arthritis of the feet or ankles.
4. Subject has a currently diagnosed progressive neurological disease such as multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, rapidly progressive arachnoiditis, brain or spinal cord tumor, or severe/critical spinal stenosis (stenosis).
5. Subjects with skin conditions in the affected dermatome that in the judgment of the investigator could interfere with evaluation of the neuropathic pain condition.
6. Subjects with other pain that may confound assessment or self-evaluation of the peripheral neuropathic pain; subjects with significant somatic pain at the site of their trauma that may confound assessment or self-evaluation of their neuropathic pain.
7. Participation in any other clinical trial within the 30 days prior to screening and/or during participation in this study.
8. Any subject considered at risk of suicide or self-harm based on investigator judgment.
9. Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormality, or other factors that may increase the risk associated with study participation or investigational product administration or may interfere with compliance or the interpretation of study results and, in the judgment of the investigator would make the subject inappropriate to participate in the study.
10. Subjects with pending Worker's Compensation, Worker's Compensation, civil litigation, or disability claims. Subjects with fully resolved litigation and compensation claims can participate.
11. Subjects who have had a diagnosis of malignancy other than basal cell carcinoma, or carcinoma in situ of the cervix within the past five years, to include life expectancy less than 1 year due to advanced malignancy.
12. Subjects with implantable "electrical" medical devices such as a cardiac pacemaker, defibrillator, or insulin pump within four (4) inches or less of the site of pain to be treated by Axon Therapy. (Subject with an implantable device greater than four (4) inches from the site of pain to be treated should NOT be excluded).
13. Phantom limb pain or pain that feels like it is coming from a body part that is no longer there.
14. Subjects who have failed other neuromodulation implantable device for the same indication
15. Subjects with shrapnel or ferromagnetic objects
16. Subject is currently taking a morphine equivalent daily dose > 120 mg/day.
17. Subject is a woman of childbearing potential, not using adequate contraception or not willing to comply with contraception for the duration of the study.
18. Subjects with active drug or alcohol abuse within 1 year prior to screening.
19. Subjects with hemoglobin A1C of 9% or higher for 90 days prior to screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Comparison of the Proportion of Responders | 30 days
  The primary efficacy endpoint is a between groups comparison of pain change from baseline to 30 days.
Comparison of therapy-related AEs between the 2 Study arms | 30 days
  The primary safety endpoint for this study is a comparison of therapy-related AEs through Day 30 between the 2 arms of the Study.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) for Pain | 30- and 90-days post-treatment
  Scores from daily diaries will be compared to baseline overall and by group (Axon therapy (AT) plus CMM and AT crossover (ATx) plus CMM)
VAS for Numbness | 30- and 90-days post-treatment
  Scores from daily diaries will be compared to baseline overall and by group (AT + CMM and ATx + CMM)
Brief Pain Inventory (BPI) | 30- and 90-days post-treatment
  Changes from baseline scores overall and by group (AT + CMM and ATx + CMM)
Daily Sleep Interference Scale (DSIS) | 30- and 90-days post-treatment
  Changes from baseline scores overall and by group (AT + CMM and ATx + CMM)
EQ-5D-3L | 30- and 90-days post-treatment
  Changes from baseline scores overall and by group (AT + CMM and ATx + CMM)
Patient Global Impression of Change (PGIC) | 30- and 90-days post-treatment
  Changes from baseline scores overall and by group (AT + CMM and ATx + CMM). In addition, the proportion of subjects with a minimal clinically important change from baseline will be compared between groups.
Depression Anxiety Stress Scales (DASS) | 30- and 90-days post-treatment
  Changes from baseline scores overall and by group (AT + CMM and ATx + CMM)
Pain Disability Index (PDI) | 30- and 90-days post-treatment
  Changes from baseline scores overall and by group (AT + CMM and ATx + CMM). In addition, the proportion of subjects with a minimal clinically important change from baseline will be compared between groups.
Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) Questionnaire | 30- and 90-days post-treatment
  Changes from baseline scores overall and by group (AT + CMM and ATx + CMM)
In-clinic VAS Pain Scores | 30- and 90-days post-treatment
  Changes from baseline scores overall and by group (AT + CMM and ATx + CMM)
Increase from baseline pain medication within four weeks of the Day 90 visit (based on prescribed doses) | 30- and 90-days post-treatment
  Changes from baseline scores overall and by group (AT + CMM and ATx + CMM)
Proportion of subjects who discontinue treatment | 30- and 90-days post-treatment
  Proportion of subjects who discontinue treatment will be compared between groups
Neurological Exam - percentage of treatment arm with a change in neurological status | 90 days post-treatment
  Percentage of treatment arm (including crossover subjects) with a change in neurological status as determined by neurological exam on Day 90 after start of active treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Milkovits, Study Director — NeuraLace Medical
Locations (7):
- United States (7):
  - Florida Pain Management Associates, P.A., Sebastian, Florida
  - Truwell Health, St. Petersburg, Florida
  - Florida Pain Management Associates, P.A., Vero Beach, Florida
  - Centurion Spine and Pain Centers, Brunswick, Georgia
  - Centurion Spine and Pain Centers, Waycross, Georgia
  - Carolinas Pain Institute and Center for Clinical Research, Winston-Salem, North Carolina
  - SC Pain and Spine Specialists, LLC, Murrells Inlet, South Carolina

REFERENCES:
- [Derived] Brown L, Gage E, Cordner H, Kapural L, Rosenberg J, Bedder M. Safety and Efficacy of Magnetic Peripheral Nerve Stimulation for Treating Painful Diabetic Neuropathy. Neuromodulation. 2025 Dec;28(8):1366-1373. doi: 10.1016/j.neurom.2025.03.074. Epub 2025 Apr 30. PMID 40304652